CLINICAL TRIAL: NCT00004113
Title: A Phase II Study of Temozolomide (SCH 52365, Temodal(R)) for the Treatment of Recurrent Malignant Glioma
Brief Title: Temozolomide in Treating Patients With Recurrent Malignant Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 99-019; CDR0000067337 (Registry Identifier: PDQ (Physician Data Query)); NCI-G99-1602
Record Dates: First submitted 1999-12-10; First posted 2004-05-21 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult glioblastoma; adult anaplastic astrocytoma; adult anaplastic oligodendroglioma; adult mixed glioma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioblastoma; Astrocytoma; Oligodendroglioma; Glioma; Gliosarcoma | interventions — Temozolomide

INTERVENTIONS:
Drug: temozolomide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of temozolomide in treating patients who have recurrent malignant glioma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety and efficacy of temozolomide in patients with recurrent malignant glioma. II. Determine the radiographic response to this regimen in these patients. III. Determine the time to tumor progression of these patients on this regimen. IV. Determine the quality of life of these patients.

OUTLINE: Patients receive oral temozolomide once daily for 42 days. Courses repeat every 70 days for up to 1 year in the absence of disease progression or unacceptable toxicity. Quality of life is assessed every 1-2 months. Patients are followed every 3-4 months.

PROJECTED ACCRUAL: A total of 20-35 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed recurrent malignant glioma, including: Glioblastoma Gliosarcoma High grade glioma Anaplastic astrocytoma Anaplastic mixed oligoastrocytoma Anaplastic oligodendroglioma Must have evidence of tumor recurrence or progression on gadolinium enhanced MRI or CT scan following radiotherapy with or without chemotherapy

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 60-100% Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 10 g/dL Hepatic: Bilirubin less than 1.5 times upper limit of normal (ULN) SGOT and SGPT less than 3 times ULN Alkaline phosphatase less than 2 times ULN Renal: Creatinine less than 1.5 times ULN BUN less than 1.5 times ULN Other: No nonmalignant systemic disease that would cause patient to be a poor medical risk No acute infection requiring intravenous antibiotics No psychological disorder that would interfere with study compliance HIV negative No AIDS-related illness Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No frequent vomiting or medical condition that would interfere with oral medication intake (e.g., partial bowel obstruction) No prior or concurrent malignancy, except: Surgically cured carcinoma in situ of the cervix Basal or squamous cell skin cancer

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior immunotherapy At least 4 weeks since prior biologic therapy Chemotherapy: See Disease Characteristics At least 4 weeks since prior chemotherapy No prior temozolomide or dacarbazine Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics At least 4 weeks since prior external beam radiotherapy At least 8 weeks since prior stereotactic radiosurgery Surgery: At least 2 weeks since prior brain biopsy, craniotomy, or other surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-06; Primary Completion 2001-10 (Actual); Study Completion 2001-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren E. Abrey, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Khan RB, Raizer JJ, Malkin MG, Bazylewicz KA, Abrey LE. A phase II study of extended low-dose temozolomide in recurrent malignant gliomas. Neuro Oncol. 2002 Jan;4(1):39-43. doi: 10.1093/neuonc/4.1.39. PMID 11772431